CLINICAL TRIAL: NCT07140939
Title: A Phase 3, Randomized, Double-blinded, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of CBL-514 Injection for Reducing Abdominal Subcutaneous Fat.
Brief Title: A Study to Evaluate the Efficacy and Safety of CBL-514 Injection for Reducing Subcutaneous Fat
Acronym: SUPREME-01
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBL-0301
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Subcutaneous Fat
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBL-514 injection (Experimental): Participants will receive CBL-514 administrated up to 120 mL (with 50 injections) per treatment at a 3-weeks interval for up to 4 treatments.
  Interventions: Drug: CBL-514 Injection
- Injectable 0.9% Sodium Chloride solution (Placebo Comparator): Participants will receive 0.9% Sodium Chloride administrated up to 120 mL (with 50 injections) per treatment at a 3-week interval for up to 4 treatments.
  Interventions: Other: 0.9% Sodium Chloride

INTERVENTIONS:
Drug: CBL-514 Injection — Provided as a ready for use injectable CBL-514 solution
  Arms: CBL-514 injection
Other: 0.9% Sodium Chloride — Injectable 0.9% Sodium Chloride solution as placebo
  Arms: Injectable 0.9% Sodium Chloride solution

SUMMARY:
A phase 3, randomized, double-blinded, placebo-controlled study to evaluate the efficacy, safety, and tolerability of CBL-514 injection for reducing abdominal subcutaneous fat.

DETAILED DESCRIPTION:
A total of approximately 300 adult participants with moderate or severe abdominal fat at Baseline 1 will be enrolled. Each participant will receive up to 4 treatments of allocated study drug administered subcutaneously to the abdomen, once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years old.
2. Body mass index (BMI) > 18.5 and < 30 kg/m2 and body weight ≥ 50 kg.
3. Participant has moderate or severe abdominal fat as assessed by the Investigator on the CR-AFRS and by the participant on the PR-AFRS.
4. Participant maintained a stable lifestyle.
5. Voluntarily signs the Informed Consent Form and is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria

1. Female participant of childbearing potential who is not willing to commit to an acceptable contraceptive method, or who is currently pregnant or lactating. Male participant who is not committing to using condom consistently and refraining from sperm donation.
2. Participant who has impeded coagulation or platelet aggregation.
3. Participant has delayed wound healing or poorly controlled diabetes.
4. Participant has active malignancies or is currently being evaluated for a possible malignancy.
5. Participant has a history of trypanophobia, the extreme fear of medical procedures involving injections or needles, or who experiences vasovagal syncope and faints at the sight of blood or a needle.
6. Participant has a visible Panniculus on the abdomen in standing position.
7. Participant has severe abdominal visceral fat.
8. Participant has skin conditions, which would pose risk to the participant if receiving the IP or interfere with the safety or efficacy evaluation.
9. Participant has undergone the procedures at the treatment area that may affect IP administration.
10. Participant with contraindications to MRI imaging.
11. Participant is on prescription or over-the-counter weight reduction medication, weight reduction programs, or taking oral or injectable GLP-1 agonists.
12. Participant is undergoing long-term systemic steroid or immunosuppressive therapy which may affect the treatment area.
13. Participant is taking or will take any medication that is known strong inhibitor or inducer of CYP1A2 enzymes, sensitive CYP1A2 substrates, or medication with narrow therapeutic index.
14. Participant with history of hypersensitivity to local anesthesia.
15. Participant with known allergies or significant adverse reaction to the IP.
16. Participant with liver cirrhosis or abnormal liver function, or with any hepatic condition that interferes with the safety or efficacy assessments.
17. Participant with any renal impairment.
18. Participant has received any investigational product.
19. Participant considered to be unreliable or incapable of complying with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with at least 13% abdominal fat change and at least a 2-grade improvement on Patient Reported Abdominal Fat Rating Scale (PR-AFRS) in the CBL-514 group versus the placebo group. | From baseline to 4 weeks after final treatment
  Measured by MRI and a 5-point ordinal scale

SECONDARY OUTCOMES:
Percentage change from baseline in abdominal fat in the CBL-514 group versus the placebo group. | From baseline to 4 weeks after final treatment
  Measured by MRI
Percentage of participants with at least a 1-grade improvement on both Participant Reported Abdominal Fat Rating Scale (PR-AFRS) and Clinician Reported Abdominal Fat Rating Scale (CR-AFRS) in the CBL-514 group versus the placebo group. | From baseline to 4 weeks after final treatment
  Measured by 5-point ordinal scales

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sheu, Study Director — Caliway Biopharmaceuticals Co., Ltd.
Locations (13):
- United States (11):
  - Investigational site 1, Encinitas, California
  - Investigational site 2, West Palm Beach, Florida
  - Investigational site 3, Chicago, Illinois
  - Investigational site 4, Baton Rouge, Louisiana
  - Investigational site 5, Hunt Valley, Maryland
  - Investigational site 6, Omaha, Nebraska
  - Investigational site 7, Hackensack, New Jersey
  - Investigational site 8, New York, New York
  - Investigational site 9, Charlotte, North Carolina
  - Investigational site 10, Nashville, Tennessee
  - Investigational site 11, Pflugerville, Texas
- Canada (2):
  - Investigational site 12, Vancouver, British Columbia
  - Investigational site 13, Toronto, Ontario